CLINICAL TRIAL: NCT01158287
Title: Phase II Study of Single Agent Sorafenib in the Treatment of Relapsed Esophageal/Gastric Adenocarcinoma in Platinum Pre-Treated Patients
Brief Title: Sorafenib. ICORG 06-41, V4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-41 ICORG; ICORG-06-41; EUDRACT-2008-005062-31; EU-21045
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-01

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: adenocarcinoma of the esophagus; recurrent esophageal cancer; recurrent gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Sorafenib

ARMS (1):
- Sorafenib 400mg bd, p.o, continuously (Experimental)
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sorafenib tosylate works in treating patients with relapsed esophageal cancer and/or stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the disease control rate (complete response, partial response, and stable disease) of sorafenib tosylate after 4 months in patients with relapsed esophageal or gastric adenocarcinoma previously treated with platinum-based chemotherapy.

Secondary

* To determine the progression-free survival of patients treated with this drug.
* To determine the overall survival of patients treated with this drug.
* To determine the time to tumor progression in patients treated with this drug.
* To determine the objective response rate in patients treated with this drug.
* To determine the tolerability and toxicity in patients treated with this drug.
* To assess biomarkers associated with response/resistance to therapy. (exploratory)

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib tosylate twice a day on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Blood and tumor samples may be collected periodically and analyzed for biological markers.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal and/or gastric adenocarcinoma

  * Relapsed or progressed disease after prior platinum-based chemotherapy and not a suitable candidate for radical therapy
* At least 1 unidimensionally measurable lesion as assessed by RECIST criteria
* No uncontrolled, symptomatic brain metastases

  * Patients with intracranial bleeding into metastases allowed provided the disease is well-controlled and not undergoing acute steroid therapy or taper (chronic steroid therapy allowed provided the dose is stable for 1 month prior to and following screening radiographic studies)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 2 months
* Hemoglobin ≥ 9.0 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT/AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* Alkaline phosphatase ≤ 2.5 times ULN (≤ 4 times ULN for patients with bony involvement)
* INR ≤ 1.5
* aPTT normal
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier method contraception prior to and during study therapy (men and women) and for 3 months after completion of study therapy (men)
* Not planning pregnancy within 6 months after completion of study therapy
* No history of cardiac disease, including any of the following:

  * NYHA class III-IV congestive heart failure
  * Active coronary artery disease (myocardial infarction more than 6 months prior to study entry allowed)
  * Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* No uncontrolled hypertension (systolic BP > 150 mm Hg or diastolic BP > 90 mm Hg, despite optimal medical management)
* No known HIV infection or chronic hepatitis B or C
* No active, clinically serious infections > CTCAE grade 2
* No thrombotic or embolic events (e.g., cerebrovascular accident including transient ischemic attacks within the past 6 months)
* No pulmonary hemorrhage or bleeding event > CTCAE grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event > CTCAE grade 3 within the past 4 weeks
* No serious, nonhealing wound, ulcer (apart from the tumor), or bone fracture
* No evidence or history of bleeding diathesis or coagulopathy
* No current signs or symptoms of severe progressive or uncontrolled hepatic, hematological, renal, endocrine, pulmonary, or cardiac disease
* No known or suspected allergy to sorafenib or any agent given in the course of this trial
* No previous cancer that is distinct in primary site or histology from esophago-gastric junction cancer except for carcinoma in situ of the cervix, treated basal cell carcinoma, superficial bladder tumors [Ta and Tis], or any cancer curatively treated > 3 years prior to study entry
* No concurrent cancer that is distinct in primary site or histology from esophago-gastric cancer
* No substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* No condition that impairs the patient's ability to swallow whole pills
* No malabsorption condition
* No seizure disorder requiring medication (e.g., steroids or antiepileptics)
* No familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No significant traumatic injury within the past 4 weeks

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior local radiotherapy
* At least 3 weeks since prior biologic response modifiers (e.g., G-CSF)

  * G-CSF and other hematopoietic growth factors allowed in the management of acute toxicity (e.g., febrile neutropenia) when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction
  * Concurrent chronic erythropoietin allowed provided no dose adjustment is undertaken within 2 months prior to the study or during the study
* At least 4 weeks since prior major surgery or open biopsy
* At least 4 weeks since prior and no concurrent radiotherapy

  * Prior or concurrent palliative radiotherapy to symptomatic disease sites allowed (unless the site to be irradiated is one of the target lesions used for response assessment)
* At least 4 weeks since prior and no concurrent anticancer chemotherapy, immunotherapy, or hormonal therapy (except bisphosphonates)
* At least 30 days since prior and no concurrent investigational drug therapy
* At least 5 weeks since prior and no concurrent mitomycin C or nitrosoureas
* At least 4 months since prior autologous bone marrow transplant or stem cell rescue
* No history of organ allograft
* No prior licensed or investigational tyrosine kinase inhibitor or antiangiogenic agent (e.g., sunitinib or bevacizumab)
* No prior sorafenib tosylate
* No prior licensed or investigational drug treatment that targets the RAS, VEGF, VEGFR, or EGFR pathway
* No concurrent rifampin or St. John wort
* No concurrent therapeutic anticoagulation with vitamin K antagonists (e.g., warfarin, heparins, or heparinoids)

  * Low-dose warfarin (1 mg by mouth once a day) allowed provided INR is < 1.5
  * Low-dose aspirin allowed
* No concurrent renal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Disease control rate after 4 months | After 4 months of treatment

SECONDARY OUTCOMES:
Progression-free survival | Ongoing
  Progression free survival and overall survival probabilities over time will be estimated using Kaplan-Meier plots. Their medians with their confidence intervals will be also presented.
  Progression Free Survival is measured from first treatment until the date of disease progression or death, whichever is reported first. Subjects who do not progress or die at the time of the analysis will be censored at the day of their last tumour assessment.
Overall survival | Ongoing
  Overall survival is measured from the date of first treatment to the date of the subject's death. If the subject is alive or the vital status is unknown, the date of death will be censored at the date that the subject is last known to be alive.
Time to tumor progression | Ongoing
Objective response rate | Response would be assessed by appropriate imaging (e.g. CT) every 8 weeks.
  The study has been designed to use the disease control rate at 4 months on treatment as the primary endpoint.
Tolerability and toxicity | Ongoing for duration of treatment and 30 day follow up.
  Patients would be assessed for toxicity according to NCI CTC version 3.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth O'Byrne, MD, Principal Investigator — St. James's Hospital, Ireland
Locations (8):
- Ireland (8):
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University College Hospital, Galway
  - Waterford Regional Hospital, Waterford